CLINICAL TRIAL: NCT03987347
Title: Health Condition of Cannabis Consumers in the Canadian Population: A Population-based Observational Cohort Study
Brief Title: Health Condition of Cannabis Consumers in the Canadian Population
Status: Withdrawn | Type: Observational
Why Stopped: No authorization from CLSA database scientific committee
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Other Study IDs: 2020-1830
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Cannabis Use; Old Age; Health Risk
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — People who are enrolled in the Canadian Longitudinal Study on Aging. Participants undergo repeated waves of the same standardized data collection every three years. All participants are also contacted by telephone 18 months after baseline assessment to complete the Maintaining Contact Questionnaire.

SUMMARY:
This study evaluates the health condition and its evolution with time of Cannabis consumers in the Canadian population.

DETAILED DESCRIPTION:
In Canada, legalization of recreational use is likely to have decreased the perception of risks associated with Cannabis use, and means that the reported adverse effects of Cannabis are not so important, suggesting that Cannabis may be useful for their illness as an alternative or complementary therapeutic.

More Canadian physicians prescribed Cannabis for their patients. Both Recreational and medical use of Cannabis increase and will continue to grow up in the next coming years. Regardless, the typology of Cannabis use, more information on the health condition of Cannabis consumers may be helpful for the medical prescription of Cannabis, in particular in older adults who are more at risk of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Living in Canada the last 20 years
* Being 60 years and over
* Being consumer of cannabis

Exclusion Criteria:

* Living outside Canada the last 20 years
* Have never consumed cannabis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People from Canada who were enrolled in the Canadian Longitudinal Study on Aging the last 20 years, and who have consumed different cannabis products for different reasons either recreational or medical.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Neurocognitive disorder | around 20 years
  The decrease of cognitive function changes the activities of daily living to older adults. Instrumental Activities of Daily Living Scale ( IADLs) will be used to assess independent living skills to people who are a diagnosis of mild cognitive impairment. A summary score range from 0 ( low function, dependent) to 8 ( high function, independent) will be given to each participant based on their daily activities.

SECONDARY OUTCOMES:
Depression | around 20 years
  It will be used the Centre for Epidemiologic Studies-Depression Scale (CES-D) that rates how often over the past week people experience symptoms that are associated with depression. In scoring the Center for Epidemiologic Studies Depression Scale, a value of 0,1,2,3 is assigned to a response based on the emotional feelings that the participants have.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada